CLINICAL TRIAL: NCT05362019
Title: Effects of One-to-one Service on the Continuation and Satisfaction of Combined Injectable Contraceptive Use.
Brief Title: Effects of One-to-one Service on the Continuation and Satisfaction of Contraceptive Use.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Institute for Family Planning, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021HX019
Record Dates: First submitted 2022-04-22; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Contraception Behavior; Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior | interventions — Family Planning Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): A mobile phone based "service system" developed by the research group will be used to provide one-to-one service for the intervention group.
  Interventions: Drug: Compound Norethisterone Enanthate Injection; Other: One-to-one Service
- control group (Active Comparator): Routine family planning services will be provided to the control group.
  Interventions: Drug: Compound Norethisterone Enanthate Injection; Other: Family Planning Service

INTERVENTIONS:
Drug: Compound Norethisterone Enanthate Injection — Combined injectable contraceptive use
Other: One-to-one Service — A mobile phone based "service system" will be used to pushing contraceptive knowledges, reminding injection, providing consultation on adverse reactions and ect.
  Arms: intervention group
Other: Family Planning Service — routine family planning service and contraceptive service.
  Arms: control group

SUMMARY:
This study aims to explore the impact of a mobile based one-to-one service model on improving the continuation and satisfaction of combined injectable contraceptive use, and improve the utilization and acceptability of efficient and long-term contraceptive methods.

DETAILED DESCRIPTION:
In China, due to the lack of understanding or misunderstanding of hormonal contraception by service providers and the public, the use of combined injectable contraceptive is not common. Therefore, this study aims to explore the impact of a mobile based one-to-one service model on improving the continuation and satisfaction of combined injectable contraceptive use, and improve the utilization and acceptability of efficient and long-term contraceptive methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old;
* Healthy Volunteers;
* More than 6 months after delivery and without lactation;
* No fertility intention within 6 months;
* Normal menstruation;
* No contraindications to the use of compound contraceptive methods;
* Had not used hormonal contraception in the previous three months;
* Understand the content and requirements of the project, be willing to cooperate, and have signed the informed consent form;
* Have a certian education level, and be able to use the special sanitary napkins to record menstrual volume and menstrual card.

Exclusion Criteria:

* Suffering from serious systemic diseases;
* Previous or current thrombotic disease;
* Malignant tumor of uterine organ;
* Unable to communicate normally due to disability or mental or intellectual impairment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Termination rate | 6 months
  The termination rates of the two groups were observed for 6 months.
Continuation rate | 6 months
  The continuation rates of the two groups were observed for 6 months.
Satisfaction rates | Up to 4 weeks
  The satisfaction rates of two groups after a 6 months of contraceptive use.

SECONDARY OUTCOMES:
Complaint of adverse reactions | Up to 9 months
  Complaint rates of various adverse reactions (dizziness / breast swelling / nausea) during different follow-up time.
Vaginal bleeding pattern | Up to 9 months
  Collecting the vaginal bleeding patterns (including menstrual onset time, duration, and termination time) in two phases (90 days in each phase) and amount of menstrual bleeding at 3 months of use by using a self-developed questionnarie and special sanitary pads for measurement.
Dysmenorrhea | Up to 9 months
  Dysmenorrhea will be collacted by a self-developed questionnarie (on a 10-point scale). A higher score indicated higher level of pain.
Waist and abdomen pain related to gynecology | Up to 9 months
  The pain will be collacted by a self-developed questionnarie (on a 10-point scale). A higher score indicated higher level of pain.
Sexual intercourse pain | Up to 9 months
  The pain will be collacted by a self-developed questionnarie (on a 10-point scale). A higher score indicated higher level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyan Pei, Principal Investigator — National Research Institute for Family Planning, China
Locations (8):
- China (8):
  - Qinghai People's Hospital, Xining, Qinghai
  - Qinghai Red Cross Hospital, Xining, Qinghai
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Tianjin Dongli hospital, Tianjin, Tianjin Municipality
  - Tianjin Jinnan hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University second hospital, Tianjin, Tianjin Municipality
  - Yunnan Xishuangbanna maternal and Child Health Hospital, Xishuangbanna Dai Autonomous Prefecture, Yunnan
  - Yunnan Xishuangbanna people's Hospital, Xishuangbanna Dai Autonomous Prefecture, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided